CLINICAL TRIAL: NCT06654193
Title: Allogeneic Adipose-derived Mesenchymal Stem Cells (MSC) for Acute Kidney Injury After Trauma or Burn
Brief Title: Allogeneic HB-adMSCs vs Placebo for the Treatment of Acute Kidney Injury
Acronym: AKI
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hope Biosciences LLC (Industry)
Collaborators: The University of Texas Health Science Center, Houston (Other); University of California, San Francisco (Other); University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Organization: Hope Biosciences Research Foundation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HBAKI01
Record Dates: First submitted 2024-10-15; First posted 2024-10-23 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Acute Kidney Injury
Keywords: acute kidney injury; stem cells; aki; hope biosciences
MeSH Terms: conditions — Acute Kidney Injury | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: This multicenter, prospective, randomized, double-blind, placebo controlled pragmatic Phase 1/Phase 2a clinical study will enroll severely injured trauma or burn patients who have developed Stage 2 AKI. Eligible patients will be randomized to receive Hope Biosciences (HB)-adMSCs or placebo administered within 24 hours of consent and in 3 doses, each 24 hours apart.
  The investigators will enroll 10 patients in Cohort 1, the Phase 1 safety substudy. All patients in Cohort 1 will receive active investigational product (IP).
  The investigators will enroll 60 patients in Cohort 2, the Phase 2a substudy; 30 patients will receive active IP, and 30 will receive placebo via randomization.
  The study population is trauma and burn patients admitted to participating hospitals who meet the inclusion and exclusion criteria. The study population will be reflective of the general trauma population at the participating sites.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Normal saline
  Interventions: Drug: Normal Saline
- Treatment (Experimental): Allogeneic adipose-derived HB-adMSCs
  Interventions: Drug: Allogeneic HB-adMSCs

INTERVENTIONS:
Drug: Allogeneic HB-adMSCs — Allogeneic HB-adMSCs
  Arms: Treatment
Drug: Normal Saline — Sterile Saline Solution
  Arms: Placebo

SUMMARY:
This study aims to investigate, through the collection of valid scientific evidence necessary to determine safety and effectiveness, the potential use of Allogeneic Hope Biosciences Adipose-derived Mesenchymal Stem Cells (HB-adMSCs) to prevent progression of trauma-induced Acute Kidney Injury (AKI).

DETAILED DESCRIPTION:
This trial multicenter, prospective, randomized, double-blind, placebocontrolled pragmatic Phase 1/Phase 2a clinical study aims to investigate, through the collection of valid scientific evidence necessary to determine safety and effectiveness, the potential use of adiposederived allogenic MSCs to prevent progression of trauma-induced AKI. We hypothesize that infusing a total of 3 doses of MSCs over 72 hours at 24-hour intervals starting in patients with modified KDIGO Stage 2 or 3 AKI will prove to be safe and efficacious.

Phase 1 of the study will include Cohort 1 (10 patients) and will confirm safety in this population with this cell formulation (cryopreserved and reanimated). Phase 2a of the study will include 60 patients (30 interventional, 30 placebo) and will look at duration of AKI at Stage 2 or higher (defined as proportion of patients with a duration of Stage 2 AKI more than 2 days after the start of treatment).

ELIGIBILITY:
Inclusion Criteria:

1. Between 18 and 75 years old AND
2. Diagnosed with Modified KDIGO Stage 2 AKI within the first 10 days after injury AND
3. Admitted to Intensive Care Unit or Intermediate Medical Unit AND
4. Received at least 3 units of any blood product within 6 hours of admission for trauma OR 15% or greater burn area OR any electrical burn OR any crush injury AND
5. Expected to survive at least 24 hours after diagnosis of KDIGO Stage 2 AKI AND
6. Patient or patient's Legally Authorized Representative (LAR) has voluntarily signed the informed consent.

Exclusion Criteria:

Patients are ineligible if they meet ONE OR MORE of the following:

1. Incarcerated individuals
2. Pregnant and lactating females
3. TBI deemed non-survivable by the trauma or neurosurgery attending physician
4. Hemodynamically unstable and requiring vasopressors for blood pressure support (systolic blood pressure ≥90 mmHg) during the 30-minute period prior to investigational product (IP) thawing/preparation
5. Pre-existing chronic kidney disease or acute kidney failure.
6. Pre-existing chronic liver disease.
7. Known immunodeficiency or concurrent use of potentially immunosuppressive medications at doses likely to result in an immunosuppressed status.
8. Active malignancy.
9. Known allergy to dimethyl sulfoxide or human serum albumin.
10. No available intravenous access (peripheral or central) of at least 22-gauge needle that can be utilized exclusively for IP during the time of planned infusion.
11. Clinical condition that would be anticipated to deteriorate with IV administration of 250 ml of crystalloid.
12. Known Do Not Resuscitate (DNR) prior to randomization

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of infusion-related adverse events (AEs) or serious adverse events (SAEs) | 1 year
  Incidence of treatment-related adverse events (TEAEs) will be monitored to assess the safety of the infusion product on the patients in Phase 1 of the trial.
Duration of Acute Kidney Injury (AKI) at Stage 2 | 2 days
  Proportion of patients with a duration of Stage 2 AKI more than 2 days after the start of treatment

SECONDARY OUTCOMES:
Number of patients with progression of Kidney Disease Improving Global Outcomes (KDIGO) Stage 2 AKI | 1 year
  The progression from Stage 2 to Stage 3 AKI often constitutes the initiation of renal replacement therapy (RRT), tripling of creatinine levels or creatinine > 4 mg/dL with an increase of 0.5 mg/dL, with an associated marked increase in morbidity, mortality, and cost.
Mortality at 30, 90 days and 365 days | 1 year
  Whether the patient remains alive or not at 1 month, 3 months, and 1 year
Post-injury organ dysfunction and thromboinflammation | 1 year
  Includes incidence of sepsis, acute respiratory distress syndrome (ARDS), venous thromboembolism (VTE; pulmonary embolism and deep venous thrombosis), and multiple organ failure (MOF)
Number of participants with chronic critical illness (≥14 days) | 1 year
  Determined by prolonged intensive care unit (ICU) admission (≥14 days) with evidence of ongoing organ dysfunction
Severity of complications, including incidence of sepsis, ARDS, venous thromboembolism (VTE; pulmonary embolism and deep venous thrombosis), and multiple organ failure (MOF) | 1 year
  Severity of each complication will be determined by complication-specific criteria, e.g. Berlin criteria (mild, moderate, severe)
Hospital-, ICU- and ventilator-free days | 1 year
  Defined as the number of days a patient was not in the hospital or on the ventilator or in the ICU at 30 days or hospital discharge/death
Number of patients with Recurrent AKI during the same hospitalization | 1 year
  Defined as the amount of patients who have several episodes of AKI in the same hospitalization

OTHER OUTCOMES:
Number of renal injury biomarkers altered by adipose-derived MSCs | 1 year
  8 plasma samples from enrolled patients at timepoints from the time of enrollment will be collected. The investigators hypothesize that MSC treatment would result in attenuation of dysregulated inflammation and endothelial injury will be reduced.

CONTACTS AND LOCATIONS:
Overall Officials: Charles S Cox, Jr., MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (3):
- United States (3):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California, San Francisco, San Francisco, California
  - University of Texas Health Science Center at Houston (UTHealth Houston), Houston, Texas